CLINICAL TRIAL: NCT07126184
Title: Incidence and Predictors of Recurrent Stroke in Patients With Cryptogenic Stroke Later Diagnosed With Atrial Fibrillation: A 5-Year Study From Lady Reading Hospital, Peshawar
Brief Title: Incidence and Predictors of Recurrent Stroke in Cryptogenic Stroke Patients With Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Nangarhar University (Other)
Responsible Party: Principal Investigator, Rafiullah Hotak, Doctor, Nangarhar University
Other Study IDs: Ref: No. 331/LRH/MTI
Record Dates: First submitted 2025-08-10; First posted 2025-08-17 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Cryptogenic Stroke; Atrial Fibrillation; Recurrent Ischemic Stroke
Keywords: Cryptogenic stroke; Atrial Fibrillation; Recurrent Ischemic Stroke; Ischemic stroke
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Extended Cardiac Monitoring — This observational study involved the use of standard cardiac monitoring methods to detect atrial fibrillation in patients initially diagnosed with cryptogenic ischemic stroke. Monitoring techniques included 12-lead ECG, 24-hour Holter monitoring, and implantable loop recorders (ILRs). No experimental interventions were assigned; patients received routine clinical care.

SUMMARY:
Brief Summary:

This study aimed to investigate the risk and factors that predict recurrent stroke in patients who initially had a stroke with no clear cause (called cryptogenic stroke) and were later found to have atrial fibrillation (AF), an irregular heart rhythm that can increase stroke risk. The study was conducted at Lady Reading Hospital in Peshawar, Pakistan, over five years from 2018 to 2023.

Stroke is a leading cause of death and disability worldwide. In many cases, the cause of stroke is unclear, which makes it difficult to prevent it from happening again. Atrial fibrillation is a common hidden cause of such strokes but is often hard to detect because it can occur intermittently without symptoms. Detecting AF early is important because patients with AF benefit greatly from blood-thinning medicines (anticoagulants) that reduce the risk of another stroke.

In this study, medical records of patients diagnosed with cryptogenic stroke were reviewed. Patients who were later diagnosed with atrial fibrillation within 12 months of their stroke were included. The researchers collected information about their age, gender, heart examinations, how and when AF was diagnosed, use of blood-thinning medicines, and if they had another stroke during follow-up.

The study highlights the importance of early and prolonged heart rhythm monitoring in patients with cryptogenic stroke to detect atrial fibrillation. It also stresses the need for better access to and adherence to anticoagulant therapy in resource-limited settings like Pakistan to reduce the risk of recurrent stroke and improve patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Patients initially diagnosed with cryptogenic ischemic stroke confirmed by neuroimaging and standard diagnostic evaluation.
* Patients subsequently diagnosed with atrial fibrillation within 12 months of index stroke, confirmed by ECG, 24-hour Holter monitoring, or implantable loop recorder.
* Availability of complete clinical and follow-up data.

Exclusion Criteria:

* Known history of atrial fibrillation or atrial flutter prior to the index stroke.
* Presence of structural heart diseases, valvular abnormalities, or congenital cardiac anomalies.
* Incomplete clinical or follow-up data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study includes adult patients admitted to Lady Reading Hospital with cryptogenic ischemic stroke who were later diagnosed with atrial fibrillation within 12 months. The cohort was followed for recurrent stroke and clinical outcomes over a median of 13.8 months.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Recurrent Ischemic Stroke | 5 years
  Occurrence of new ischemic stroke confirmed by clinical assessment and neuroimaging during the follow-up period in patients initially diagnosed with cryptogenic stroke and later diagnosed with atrial fibrillation.

CONTACTS AND LOCATIONS:
Locations (1):
- LRH/MTI, Peshawar, KPK, Pakistan

IPD SHARING:
Plan to Share IPD: No